CLINICAL TRIAL: NCT04850794
Title: Evaluation of an Interdisciplinary Decision Guide for Infant Feeding Assessment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Screening
Other Study IDs: 20-2786
Record Dates: First submitted 2021-04-14; First posted 2021-04-20 (Actual); Results first posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2022-03

CONDITIONS: Premature Birth; Feeding and Eating Disorders of Childhood
Keywords: early intervention; pediatric feeding; assessment
MeSH Terms: conditions — Premature Birth; Feeding and Eating Disorders of Childhood

STUDY DESIGN:
Intervention Model Description: Therapists will answer clinical questions about a case study (A or B, randomized order of presentation) without using the tool. They will then be presented with the tool and will answer the same clinical questions about a second case study (A or B, randomized order of presentation)
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case A then Case B (Experimental): Participant will first review and answer questions about Case A without using the tool. Then, they will use the tool to answer questions about case B.
  Interventions: Behavioral: Decision Support Tool
- Case B then Case A (Experimental): Participant will first review and answer questions about Case B without using the tool. Then, they will use the tool to answer questions about case A.
  Interventions: Behavioral: Decision Support Tool

INTERVENTIONS:
Behavioral: Decision Support Tool — The decision support tool is an observational checklist with recommendations for specific specialist referrals based on what the provider observed during the feeding evaluation.

SUMMARY:
Preterm infants are at risk for feeding problems which can persist through early childhood. These feeding problems may include oral motor, sensory, digestive, nutritional, respiratory, and/or behavioral components. In North Carolina's early intervention program, speech pathologists or occupational therapists are responsible for completing feeding evaluations, and may not know when to refer infants out to medical specialists to address these other domains. This study will test a decision support tool in hypothetical feeding evaluation scenarios. The hypothetical scenarios will consist of real feeding videos of preterm infants who recently participated in a multidisciplinary feeding evaluation. Parent-reported outcomes of the infant's real evaluation will be compared to those of the speech pathologists and occupational therapists in our study who do, and do not, use the decision support tool. The investigators hypothesize that therapists with the tool will make recommendations that are closer to those of the multidisciplinary team, and that they will find the tool useful and easy to use.

Due to recruitment limitations with families, the study was adapted in October, 2021 prior to enrollment of subjects to use case studies, rather than infant videos, as the hypothetical situation from which to test the tool. Therapists will then answer clinical questions without using the tool when viewing the first case study, and will use the tool to answer questions when viewing the second case study. Order of case study presentation will be randomized among participants.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age,
* speech language pathologist or occupational therapist,
* at least 2 years of experience evaluating and treating pediatric feeding,
* have worked in early intervention in last 5 years,
* English proficiency,
* currently reside in North Carolina

Exclusion Criteria:

* <2 years of experience in pediatric feeding,
* have not worked in Early Intervention in last 5 years,
* younger than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2021-07-14 (Actual); Primary Completion 2022-02-07 (Actual); Study Completion 2022-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelsey Thompson, MS, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University of North Carolina.
Time Frame: 9 to 36 months following publication
Access Criteria: The investigator who proposes to use the data has IRB, IEC, or REB approval, as applicable, and an executed data use/sharing agreement with the University of North Carolina.

REFERENCES:
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459

RESULTS

PARTICIPANT FLOW:
Period: Read 1st Case Study Without Tool
Arm/Group | Case A Then Case B | Case B Then Case A
Started | 28 | 28
Completed | 28 | 28
Not Completed | 0 | 0
Period: Read 2nd Case Study With Tool
Arm/Group | Case A Then Case B | Case B Then Case A
Started | 28 | 28
Completed | 28 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Case A Then Case B | Case B Then Case A | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age data were not collected from any participant.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 28 | 56
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28 | 28 | 56
Year of Graduation For Clinical Degree [Count of Participants; unit: Participants] — Population: One participant did not report this data.
  Participants
    number analyzed (Participants) | 28 | 27 | 55
    1980-1989 | 1 | 1 | 2
    1990-1999 | 5 | 4 | 9
    2000-2009 | 1 | 4 | 5
    2010-2019 | 21 | 18 | 39
    2020 or later | 0 | 0 | 0
Years of Pediatric Feeding Experience [Count of Participants; unit: Participants]
  2 years or less | 4 | 4 | 8
  3-5 years | 15 | 10 | 25
  6-8 years | 2 | 7 | 9
  9-11 years | 3 | 1 | 4
  12 or more years | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Recommend Feeding Therapy
Description: After reading a feeding case study, early intervention professionals will answer the question "Would you recommend feeding therapy?" with two choices: yes or no. Difference in agreement between early intervention professionals using the decision support tool and those not will be calculated and compared for cases A and B.
Time Frame: Immediately after reading feeding case study, within approximately 5 minutes
Population: Participant responses to Case A and Case B were analyzed separately.
Measure: Count of Participants; unit: Participants
Groups:
- With Decision Support Tool: Decision Support Tool: The decision support tool is an observational checklist with recommendations for specific specialist referrals based on what the provider observed during the feeding evaluation.
- Without Decision Support Tool: Unaided by Decision Support Tool
Arm/Group | With Decision Support Tool | Without Decision Support Tool
Number analyzed (Participants) | 56 | 56
Participants
  Case A-"Yes" response: number analyzed (Participants) | 28 | 28
  Case A-"Yes" response | 27 | 27
  Case A-"No" response: number analyzed (Participants) | 28 | 28
  Case A-"No" response | 1 | 1
  Case B-"Yes" response: number analyzed (Participants) | 28 | 28
  Case B-"Yes" response | 26 | 25
  Case B-"No" response: number analyzed (Participants) | 28 | 28
  Case B-"No" response | 2 | 3

2. Primary Outcome: Number of Participants That Recommend Referral to Other Providers
Description: After reading a feeding case study, early intervention professionals will answer the question "Would you refer this family to any other providers/specialists for evaluation/treatment?" with two answer choices: yes or no. Difference in agreement between early intervention professionals using the decision support tool and those not will be calculated and compared for cases A and B.
Time Frame: Immediately after reading feeding case study, within approximately 5 minutes
Population: Participant responses to Case A and Case B were analyzed separately.
Measure: Count of Participants; unit: Participants
Arm/Group | With Decision Support Tool | Without Decision Support Tool
Number analyzed (Participants) | 56 | 56
Participants
  Case A-"Yes" response: number analyzed (Participants) | 28 | 28
  Case A-"Yes" response | 27 | 25
  Case A-"No" response: number analyzed (Participants) | 28 | 28
  Case A-"No" response | 1 | 3
  Case B-"Yes" response: number analyzed (Participants) | 28 | 28
  Case B-"Yes" response | 27 | 25
  Case B-"No" response: number analyzed (Participants) | 28 | 28
  Case B-"No" response | 1 | 3

3. Primary Outcome: Number of Participants That Recommend Referral by Specialty
Description: After reading the feeding case study, early intervention professionals will answer the question "What other professionals would you refer this child to? Check all that apply." with the following choices: nutritionist/dietician, gastroenterologist, otolaryngologist (ENT), aerodigestive clinic, pulmonologist, occupational therapist, speech language pathologist, psychologist/social worker, applied behavior analyst (ABA), or allergist. Difference in agreement between early intervention professionals using the decision support tool and those not will be calculated and compared for cases A and B.
Time Frame: Immediately after reading feeding case study, within approximately 5 minutes
Population: The question was only answered by those participants who recommended referring to another professional. Participant responses to Case A and Case B were analyzed separately.
Measure: Count of Participants; unit: Participants
Arm/Group | With Decision Support Tool | Without Decision Support Tool
Number analyzed (Participants) | 54 | 50
Participants
  Case A Nutritionist/dietician: number analyzed (Participants) | 27 | 25
  Case A Nutritionist/dietician | 11 | 3
  Case A-Gastroenterologist: number analyzed (Participants) | 27 | 25
  Case A-Gastroenterologist | 20 | 17
  Case A-Otolaryngologist (ENT): number analyzed (Participants) | 27 | 25
  Case A-Otolaryngologist (ENT) | 2 | 4
  Case A-Aerodigestive clinic: number analyzed (Participants) | 27 | 25
  Case A-Aerodigestive clinic | 9 | 1
  Case A-Pulmonologist: number analyzed (Participants) | 27 | 25
  Case A-Pulmonologist | 0 | 0
  Case A-Occupational therapist and speech language pathologist: number analyzed (Participants) | 27 | 25
  Case A-Occupational therapist and speech language pathologist | 16 | 14
  Case A-Psychologist/social worker: number analyzed (Participants) | 27 | 25
  Case A-Psychologist/social worker | 1 | 0
  Case A-Applied behavior analyst (ABA): number analyzed (Participants) | 27 | 25
  Case A-Applied behavior analyst (ABA) | 1 | 0
  Case A-Allergist: number analyzed (Participants) | 27 | 25
  Case A-Allergist | 0 | 3
  Case A-Multi-disciplinary team: number analyzed (Participants) | 27 | 25
  Case A-Multi-disciplinary team | 12 | 11
  Case A-Other: number analyzed (Participants) | 27 | 25
  Case A-Other | 1 | 8
  Case B-Nutritionist/dietician: number analyzed (Participants) | 27 | 25
  Case B-Nutritionist/dietician | 10 | 8
  Case B-Gastroenterologist: number analyzed (Participants) | 27 | 25
  Case B-Gastroenterologist | 15 | 11
  Case B-Otolaryngologist (ENT): number analyzed (Participants) | 27 | 25
  Case B-Otolaryngologist (ENT) | 10 | 6
  Case B-Aerodigestive clinic: number analyzed (Participants) | 27 | 25
  Case B-Aerodigestive clinic | 15 | 4
  Case B-Pulmonologist: number analyzed (Participants) | 27 | 25
  Case B-Pulmonologist | 1 | 1
  Case B-Occupational therapist and speech language pathologist: number analyzed (Participants) | 27 | 25
  Case B-Occupational therapist and speech language pathologist | 10 | 12
  Case B-Psychologist/social worker: number analyzed (Participants) | 27 | 25
  Case B-Psychologist/social worker | 1 | 0
  Case B-Applied behavior analyst (ABA): number analyzed (Participants) | 27 | 25
  Case B-Applied behavior analyst (ABA) | 2 | 0
  Case B-Allergist: number analyzed (Participants) | 27 | 25
  Case B-Allergist | 4 | 1
  Case B-Multi-disciplinary team: number analyzed (Participants) | 27 | 25
  Case B-Multi-disciplinary team | 21 | 14
  Case B-Other: number analyzed (Participants) | 27 | 25
  Case B-Other | 6 | 7

4. Secondary Outcome: Number of Participants That Recommend Feeding Therapy Categorized by Number of Times Per Week
Description: After reading the feeding case study, early intervention professionals who recommended feeding therapy will answer the question "With what frequency would you recommend therapy?" with three choices: 2 times per week or more, 1 time per week, less than one time per week. Difference in agreement between early intervention professionals using the decision support tool and those not will be calculated and compared for cases A and B.
Time Frame: Immediately after reading feeding case study, within approximately 5 minutes
Population: The question was only answered by those participants who recommended feeding therapy. Participant responses to Case A and Case B were analyzed separately.
Measure: Count of Participants; unit: Participants
Arm/Group | With Decision Support Tool | Without Decision Support Tool
Number analyzed (Participants) | 53 | 52
Participants
  Case A-2 times per week or more: number analyzed (Participants) | 27 | 27
  Case A-2 times per week or more | 8 | 3
  Case A-1 time per week: number analyzed (Participants) | 27 | 27
  Case A-1 time per week | 19 | 24
  Case A-less than one time per week: number analyzed (Participants) | 27 | 27
  Case A-less than one time per week | 0 | 0
  Case B-2 times per week or more: number analyzed (Participants) | 26 | 25
  Case B-2 times per week or more | 12 | 13
  Case B-1 time per week: number analyzed (Participants) | 26 | 25
  Case B-1 time per week | 14 | 12
  Case B-less than one time per week: number analyzed (Participants) | 26 | 25
  Case B-less than one time per week | 0 | 0

5. Secondary Outcome: Number of Participants That Recommend Intervention Target Choices
Description: After reading the feeding case study, early intervention professionals who recommended feeding therapy will answer the question "What therapy targets might you include for this child?" and may check all that apply from the following choices: oral motor skills, sensory, behavioral, medication, modification of food/liquid, modification of equipment (seating, utensils, etc.), modification of environment (location, distractions, routine, etc.), parent coaching, or other. Difference in agreement between early intervention professionals using the decision support tool and those not will be calculated and compared for cases A and B.
Time Frame: Immediately after reading feeding case study, within approximately 5 minutes
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | With Decision Support Tool | Without Decision Support Tool
Number analyzed (Participants) | 53 | 52
Participants
  Case A-Oral Motor Skills: number analyzed (Participants) | 27 | 27
  Case A-Oral Motor Skills | 26 | 25
  Case A-Sensory: number analyzed (Participants) | 27 | 27
  Case A-Sensory | 22 | 19
  Case A-Behavioral: number analyzed (Participants) | 27 | 27
  Case A-Behavioral | 22 | 11
  Case A-Medication: number analyzed (Participants) | 27 | 27
  Case A-Medication | 4 | 5
  Case A-Modification of food/liquid: number analyzed (Participants) | 27 | 27
  Case A-Modification of food/liquid | 15 | 16
  Case A-Modification of Equipment: number analyzed (Participants) | 27 | 27
  Case A-Modification of Equipment | 12 | 8
  Case A-Modification of Environment: number analyzed (Participants) | 27 | 27
  Case A-Modification of Environment | 16 | 14
  Case A-Parent Coaching: number analyzed (Participants) | 27 | 27
  Case A-Parent Coaching | 27 | 27
  Case A-Other: number analyzed (Participants) | 27 | 27
  Case A-Other | 2 | 3
  Case B-Oral Motor Skills: number analyzed (Participants) | 26 | 25
  Case B-Oral Motor Skills | 26 | 23
  Case B-Sensory: number analyzed (Participants) | 26 | 25
  Case B-Sensory | 11 | 9
  Case B-Behavioral: number analyzed (Participants) | 26 | 25
  Case B-Behavioral | 6 | 1
  Case B-Medication: number analyzed (Participants) | 26 | 25
  Case B-Medication | 2 | 0
  Case B-Modification of food/liquid: number analyzed (Participants) | 26 | 25
  Case B-Modification of food/liquid | 22 | 24
  Case B-Modification of Equipment: number analyzed (Participants) | 26 | 25
  Case B-Modification of Equipment | 26 | 24
  Case B-Modification of Environment: number analyzed (Participants) | 26 | 25
  Case B-Modification of Environment | 24 | 21
  Case B-Parent Coaching: number analyzed (Participants) | 26 | 25
  Case B-Parent Coaching | 26 | 25
  Case B-Other: number analyzed (Participants) | 26 | 25
  Case B-Other | 3 | 4

6. Secondary Outcome: Decision Support Tool Acceptability Score
Description: The Acceptability of Intervention Measure (AIM) will be used to measure acceptability of the decision support tool. This tool includes four items, rated on a five-point Likert scale from completely disagree to completely agree, and will be quantified with a score of 0 for completely disagree, 1 for disagree, 2 for neither agree nor disagree, 3 for agree, and 4 for completely agree. The average score across the four items will be calculated, with higher scores indicating higher acceptability of the decision making tool. The minimum score is 0 and the maximum score is 4. Items on this measure include: (Intervention) meets my approval; (Intervention) is appealing to me; I like (Intervention) and I welcome (Intervention).
Time Frame: Immediately after using tool, within approximately 5 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- All Participants: Includes all participants who used the Decision Support Tool
Arm/Group | All Participants
Number analyzed (Participants) | 56
score on a scale | 3.40 (0.52)

7. Secondary Outcome: Decision Support Tool Appropriateness Score.
Description: The Intervention Appropriateness Measure (IAM) will be used to measure appropriateness of the decision support tool. This tool includes four items, rated on a five-point Likert scale from completely disagree to completely agree, and will be quantified with a score of 0 for completely disagree, 1 for disagree, 2 for neither agree nor disagree, 3 for agree, and 4 for completely agree. The average score across the four items will be calculated, with higher scores indicating higher acceptability of the decision making tool. The minimum score is 0 and the maximum score is 4. Items on this measure include: (Intervention) seems fitting; (Intervention) seems suitable; (Intervention) seems applicable; (Intervention) seems like a good match.
Time Frame: Immediately after using tool, within approximately 5 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 56
score on a scale | 3.37 (0.54)

8. Secondary Outcome: Decision Support Tool Feasibility Score.
Description: The Feasibility of Intervention Measure (FIM) will be used to measure feasibility of use of the decision support tool. This tool includes four items, rated on a five-point Likert scale from completely disagree to completely agree, and will be quantified with a score of 0 for completely disagree, 1 for disagree, 2 for neither agree nor disagree, 3 for agree, and 4 for completely agree. The average score across the four items will be calculated, with higher scores indicating higher acceptability of the decision making tool. The minimum score is 0 and the maximum score is 4. Items on this measure include: (Intervention) seems implementable; (Intervention) seems possible; (Intervention) seems doable; (Intervention) seems easy to use.
Time Frame: Immediately after using tool, within approximately 5 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 56
score on a scale | 3.50 (0.57)

ADVERSE EVENTS:
Time Frame: From the time of signing the informed consent through survey completion, an average of 10 minutes.
Description: Provider responses were monitored weekly for any concerning responses for this survey study.
Groups:
- Case A With Decision Support Tool; Case B With Decision Support Tool: Decision Support Tool: The decision support tool is an observational checklist with recommendations for specific specialist referrals based on what the provider observed during the feeding evaluation.
- Case A Without Decision Support Tool; Case B Without Decision Support Tool: Unaided by Decision Support Tool
Arm/Group | Case A With Decision Support Tool | Case B With Decision Support Tool | Case A Without Decision Support Tool | Case B Without Decision Support Tool
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28 | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28 | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28 | 0/28 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-18): https://cdn.clinicaltrials.gov/large-docs/94/NCT04850794/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-18): https://cdn.clinicaltrials.gov/large-docs/94/NCT04850794/ICF_001.pdf